CLINICAL TRIAL: NCT07251894
Title: HF-MTM Pilot: Pilot Study Exploring the Feasibility, Acceptability, and Impact of Medically Tailored Meals on Post-Discharge Recovery in Patients With Heart Failure
Brief Title: Pilot Study Exploring the Feasibility, Acceptability, and Impact of Medically Tailored Meals on Post-Discharge Recovery in Patients With Heart Failure
Acronym: HF-MTM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 859165
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Medically tailored meals; Food is medicine; Food as medicine; Heart failure; Diet quality; Readmissions
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medically Tailored Meals (Experimental): Participants can choose to receive a weekly delivery of 7, 14, or 21 medically tailored meals at no cost to them for 4 weeks.
  Interventions: Other: Medically Tailored Meals

INTERVENTIONS:
Other: Medically Tailored Meals — Medically tailored meals to provide essential tailored nutrition for patients recovering from a heart failure hospitalization

SUMMARY:
The goal of this interventional pilot study is to evaluate the feasibility, acceptability, and impact of medically tailored meals (MTM) on post-discharge recovery in patients with heart failure for Penn Medicine patients in Philadelphia and Lancaster through two pilots.

DETAILED DESCRIPTION:
Pilot 1: Will enroll 30 eligible Penn Medicine patients to receive 4 weeks of medically tailored meals (MTMs) directly to their door. Patients will be given the opportunity to choose to receive 7/14/21 meals from the MTM provider for the duration of their participation in the 4 week pilot.

Pilot 1 participants will be asked to complete a baseline survey, and end of study survey, and an end of study semi-structured interview.

Pilot 2: Will expand upon the learnings from Pilot 1 and be a larger scale longer Food is Medicine (FIM) intervention with patients receiving 8 weeks of MTM deliveries directly to their door. As with Pilot 1, patients will be given the opportunity to choose to receive 7/14/21 meals from the MTM provider for the duration of their participation in the 8 week pilot.

Pilot 2 participants will be asked to complete a baseline survey, a mid-point survey at 4 weeks, and an end of study survey and semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Have a primary diagnosis of health failure based on ICD code I50* with active hospitalization at time of enrollment
* Must be insured by Medicaid or Medicare or dual eligible
* Ability to read and speak English
* Ability to provide informed consent

Exclusion Criteria:

* Are on hospice care or reside in an acute or skilled nursing facility
* Are undergoing evaluation for advanced HF treatments including heart transplant or ventricular assist devices
* Are unable to complete data collection due to cognitive decline or disability (based on the electronic health record or referring provider assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the MTM intervention | From enrollment to the end of the intervention at 4 weeks for Pilot 1
  The % of meals successfully delivered to the patient, where a 75% rate of successful delivery indicates feasibility.
Acceptability of the MTM intervention as measured by the Net Promoter Score | At the end of the intervention at 4 weeks for Pilot 1.
  Will evaluate the acceptability of the intervention among patients through the Net Promoter Score (scale of 0 to 10; 9-10 being promoters, 7-8 being passives, and 0-6 being detractors)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States